CLINICAL TRIAL: NCT01248585
Title: A Randomized Phase III Double-Blind Study of Dexamethasone Versus Placebo in the Prophylaxis of Radiation-Induced Pain Flare Following Palliative Radiotherapy for Bone Metastases
Brief Title: Dexamethasone vs Placebo in the Prophylaxis of Radiation-Induced Pain Flare Following Palliative Radiotherapy for Bone Metastases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SC23
Record Dates: First submitted 2010-11-22; First posted 2010-11-25 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2020-04

CONDITIONS: Bone Metastases
Keywords: Symptom Control
MeSH Terms: interventions — Dexamethasone; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Active Comparator): 2 x 4 mg dexamethasone tablets taken once daily for 5 days
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): 2 placebo tablets taken once daily for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — 2 x 4 mg dexamethasone (dex) tablets taken once daily for 5 days
  Arms: Dexamethasone
Drug: Placebo — 2 placebo tablets taken once daily for 5 days
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
This research is being done because is is not known if dexamethasone can prevent pain flare (their pain temporarily gets worse before it gets better) caused by the radiation used to treat painful bone metastases. Using dexamethasone to prevent pain like this has been studied in a few people and seems promising, but it is not clear if it can decrease the pain or prevent the pain flare before it happens.

DETAILED DESCRIPTION:
Previous research has shown that for patients who receive radiation therapy to treat their painful bone metastases, about 2 out of every 5 patients (about 40%) experience pain flare. The purpose of this study is to find out whether pain flare is prevented by receiving 8mg dexamethasone at least one hour prior to radiotherapy and once daily for the following 4 days. To do this, half of the patients in this study will get dexamethasone and the other half will receive a placebo (a substance that does not do anything). Using a placebo is the best way to see if a new therapy is effective and to clearly see the potential side effects and impact on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Have a histologically or cytologically proven malignancy. All non-hematologic malignant tumours of any histology are eligible.
* Be 18 years of age or older at the time of randomization.
* Have bone metastasis(es) corresponding to the clinically painful area(s) documented by radiological imaging within six months prior to randomization.
* Karnofsky Performance Status (KPS) must be ≥ 40 at the time of the baseline evaluation (within seven days prior to randomization). As it is difficult to obtain complete data from inpatients on a daily basis, they should not be randomized to this study.
* Is planned to receive palliative radiotherapy to one or two bony metastasis(es) with the treatment given as 8 Gy in a single fraction to all sites to be followed for the study. Although a maximum of two sites can be treated and followed for the study, patients with more than two skeletal metastases are eligible. At the time of delivery of study radiotherapy, only the site(s) being followed for the study may be treated.
* Is able to provide the worst pain score at the bony metastatic site(s) planned for palliative radiotherapy.
* Has a baseline worst pain score ≥ 2 on a scale of 0-10 at all the bony metastatic site(s) planned for palliative radiotherapy as part of this study within 7 days prior to randomization. If two painful sites will be followed for the study, this requirement must be met on the same day for both sites.
* Is able and willing to fill out the daily diary.
* Is able (i.e. sufficiently fluent) and willing to complete the quality of life questionnaire in either English or French. The baseline assessment must be completed within required timelines prior to randomization. Inability (illiteracy in English or French, loss of sight, or other equivalent reason) to complete the questionnaires will not make the patient ineligible for the study. However, ability but unwillingness to complete the questionnaires will make the patient ineligible.
* Patient consent must be obtained according to local Institutional and/or University Human Experimentation Committee requirements. It will be the responsibility of the local participating investigators to obtain the necessary local clearance, and to indicate in writing to the NCIC CTG Study Coordinator that such clearance has been obtained, before the trial can commence in that centre. Because of differing requirements, a standard consent form for the trial will not be provided but a sample form is provided. A copy of the initial full board REB approval and approved consent form must be sent to the central office. The patient must sign the consent form prior to randomization. Please note that the consent form for this study must contain a statement which gives permission for the NCIC CTG and monitoring agencies to review patient records.
* If being enrolled through a centre participating in the correlative science component of the study, is willing and able to provide a pre- and post-treatment urine sample. Language pertaining to patient consent for urine collection must be included in the consent form for the main study at these centres. The patient must sign this consent form prior to collection of the first urine sample.
* If being enrolled through a centre participating in the correlative science component of the study, patient consent for the saliva collection component of the trial must be obtained in the same manner as outlined above for the main study consent. The patient must sign the saliva collection Informed Consent form.
* Must be accessible for treatment and follow-up. Investigators must be reasonably assured that the patients randomized on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.
* Protocol treatment is to begin within one week of patient randomization.

Exclusion Criteria:

* Patients with hematologic malignancies (leukemia, Hodgkin's or non-Hodgkin's lymphoma or plasma cell dyscrasia, including multiple myeloma) are ineligible as steroids constitute anti-cancer therapy for these malignancies.
* Concurrent use or use within previous seven days of any corticosteroid medication other than topical or inhaled preparations. Patients with any type of cancer who are receiving steroids as a component of their systemic therapy are ineligible. Patients requiring steroids for a co-existing medical problem are ineligible. Patients who received a one- to three-day dose of steroids as an antiemetic for chemotherapy treatment are eligible, as long as at least 72 hours have elapsed since the last dose of antiemetic therapy.
* Medical contraindications to corticosteroids such as uncontrolled diabetes mellitus, uncontrolled hypertension, active peptic ulcer or hypokalemia.
* Uncorrected hypokalemia that is known to exist within 7 days prior to randomization. Patients with previous hypokalemia that has been corrected are eligible. Hypokalemia is defined as a potassium level < 3.0 mmol/L. Testing of electrolytes, including potassium level, is not a protocol requirement.
* Random glucose level ≥ 13.9 mmol/L within 7 days prior to randomization.Testing of glucose within 7 days prior to randomization is a protocol requirement. Point of care testing with a glucometer is permissible.
* Pathological fracture of the femora, tibiae, fibulae, humeri, radii or ulnae at the site(s) to be followed for the study.
* Radiological evidence of high-risk lesions for pathological fractures in the femora, tibiae, fibulae, humeri, radii or ulnae at the site(s) to be followed for the study (lytic lesions > 3 cm or > 50% cortical erosion of bone diameter).
* Clinical or available radiologic evidence of spinal cord or cauda equina compression at the site(s) to be followed for the study.
* Plans to receive palliative radiotherapy to a site or sites other than the one(s) being followed for the study during the ten-day period following study radiotherapy.
* Planned orthopedic intervention, including kyphoplasty, vertebroplasty or cementoplasty, to any of the site(s) to be followed for the study.
* Prior palliative surgery to any of the site(s) to be followed for the study.
* Inability, with available translator assistance, to record pain score and medication consumption in the daily diary and to communicate this to study personnel.
* Receipt of radiopharmaceutical treatment at any time.
* Previous external beam radiotherapy (including hemibody radiotherapy) using a field that included the site(s) to be followed for the study.
* Inability to swallow or tolerate oral medications, e.g. due to intractable nausea and/or emesis.
* Plans to receive cytotoxic chemotherapy or systemic steroids during the on-study period (day of study radiotherapy and the subsequent ten days).
* Plans to start or stop systemic therapy other than cytotoxic chemotherapy (e.g. hormonal therapy; immunotherapy; bisphosphonates) during the on-study period (day of study radiotherapy and the subsequent ten days). Patients who are already receiving these types of treatments are eligible as long as no changes are planned during the study period.
* Regular use of a non-steroidal anti-inflammatory drug (NSAID). Patients must not be taking NSAIDs at randomization and their use during the on-study period (day of study radiotherapy and the subsequent ten days) must not be required or expected. Patients who use daily low-dose ASA for anti-platelet therapy are eligible if ASA has been used for more than one month prior to the time of randomization.
* Plans for a change in analgesic regimen on the day of randomization.
* Previous entry on the SC.23 study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2011-05-30 (Actual); Primary Completion 2015-05-25 (Actual); Study Completion 2015-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward LW Chow, Study Chair — Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto ON; Carlo De Angelis, Study Chair — Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto ON; Alysa Fairchild, Study Chair — Cross Cancer Institute, Edmonton AB
Locations (22):
- Canada (22):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Abbotsford Centre, Abbotsford, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - BCCA - Vancouver Island Cancer Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Vitalite Health Network - Dr. Leon Richard, Moncton, New Brunswick
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - London Regional Cancer Program, London, Ontario
  - Stronach Regional Health Centre at Southlake, Newmarket, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - CHUQ-Pavillon Hotel-Dieu de Quebec, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chow E, Meyer RM, Ding K, Nabid A, Chabot P, Wong P, Ahmed S, Kuk J, Dar AR, Mahmud A, Fairchild A, Wilson CF, Wu JSY, Dennis K, Brundage M, DeAngelis C, Wong RKS. Dexamethasone in the prophylaxis of radiation-induced pain flare after palliative radiotherapy for bone metastases: a double-blind, randomised placebo-controlled, phase 3 trial. Lancet Oncol. 2015 Nov;16(15):1463-1472. doi: 10.1016/S1470-2045(15)00199-0. Epub 2015 Oct 18. PMID 26489389
- [Derived] Chow S, Ding K, Wan BA, Brundage M, Meyer RM, Nabid A, Chabot P, Coulombe G, Ahmed S, Kuk J, Dar AR, Mahmud A, Fairchild A, Wilson CF, Wu JSY, Dennis K, DeAngelis C, Wong RKS, Zhu L, Chow E. Gender differences in pain and patient reported outcomes: a secondary analysis of the NCIC CTG SC. 23 randomized trial. Ann Palliat Med. 2017 Dec;6(Suppl 2):S185-S194. doi: 10.21037/apm.2017.08.12. Epub 2017 Aug 29. PMID 29156903
- [Derived] McDonald R, Ding K, Brundage M, Meyer RM, Nabid A, Chabot P, Coulombe G, Ahmed S, Kuk J, Dar AR, Mahmud A, Fairchild A, Wilson CF, Wu JSY, Dennis K, DeAngelis C, Wong RKS, Zhu L, Chan S, Chow E. Effect of Radiotherapy on Painful Bone Metastases: A Secondary Analysis of the NCIC Clinical Trials Group Symptom Control Trial SC.23. JAMA Oncol. 2017 Jul 1;3(7):953-959. doi: 10.1001/jamaoncol.2016.6770. PMID 28196208
- [Derived] Raman S, Ding K, Chow E, Meyer RM, Nabid A, Chabot P, Coulombe G, Ahmed S, Kuk J, Dar AR, Mahmud A, Fairchild A, Wilson CF, Wu JSY, Dennis K, DeAngelis C, Wong RKS, Zhu L, Brundage M. Minimal clinically important differences in the EORTC QLQ-BM22 and EORTC QLQ-C15-PAL modules in patients with bone metastases undergoing palliative radiotherapy. Qual Life Res. 2016 Oct;25(10):2535-2541. doi: 10.1007/s11136-016-1308-4. Epub 2016 May 2. PMID 27138964

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexamethasone | Placebo
Started | 148 | 150
Completed | 148 | 150
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: ITT
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone | Placebo | Total
Number analyzed (Participants) | 148 | 150 | 298
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (12.9) | 68.6 (12) | 67.6 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 68 | 128
  Male | 88 | 82 | 170
Region of Enrollment [Number; unit: participants]
  Canada | 148 | 150 | 298
Primary cancer site [Number; unit: participants]
  Breast | 33 | 33 | 66
  Lung | 41 | 39 | 80
  Prostate | 36 | 38 | 74
  Others | 38 | 40 | 78
Number of painful sites [Number; unit: participants]
  1 | 115 | 116 | 231
  2 | 33 | 34 | 67

OUTCOME MEASURES:

1. Primary Outcome: Radiation-induced Pain Flare Incidence
Description: The incidences of radiation-induced pain flare from the time of radiotherapy treatment to ten days after the completion of treatment
Time Frame: 10 days
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 148 | 150
Participants | 39 | 53
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; One-sided 0.05 level test with 90% power, 298 participants required; Test type: Superiority; p = 0.05, Cochran-Mantel-Haenszel — 1-sided p-value; Risk Difference (RD) = 0.09, 90% CI 2-sided [0 to 0.177], Standard Error of Mean 0.053

2. Secondary Outcome: Radiation-induced Pain Flare Incidence From Day 6 to Day 10 After Radiotherapy Treatment
Description: Reduction in incidence of radiation-induced pain flare from Day 6 to Day 10 after radiotherapy treatment
Time Frame: From Day 6 to day 10 after radiotherapy treatment
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 148 | 150
Participants | 32 | 35
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Test type: Superiority or Other; p = 0.432, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.009, 95% CI 2-sided [-0.08 to 0.10]

3. Secondary Outcome: Analgesic Use
Description: Change in mean analgesic use from baseline to day 10.
Time Frame: 10 days
Population: Patients with baseline and day 10 Analgesic Use data.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 126 | 129
mg | 1.29 (36.0) | 9.83 (59.4)

4. Secondary Outcome: Response to Radiation Treatment at Six Weeks
Description: Response to radiation treatment at six weeks after treatment. Complete response (CR) is defined as a worst pain score of zero (0) at the bony metastatic site with no concomitant increase in analgesic intake (stable or reduced oral morphine equivalent dosage (OMED)).
  Partial response (PR) is defined as any of the following:
  i. Reduction in worst pain score of two or more at the bony metastatic site on a 0-10 scale without analgesic increase.
  ii. Analgesic reduction of 25% or more from baseline without an increase in worst pain score with reference to baseline.
  iii. For patients who were using opioid analgesics at the baseline assessment, a daily oral morphine equivalence of zero (0) without an increase in worst pain score relative to the baseline worst pain score
Time Frame: From day 0 to 6 weeks
Population: ITT
Measure: Number; unit: participants
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 148 | 150
participants | 64 | 52
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Test type: Superiority; p = 0.15, Fisher Exact — Fisher exact test; Risk Difference (RD) = 0.09, 90% CI 2-sided [0.01 to 0.18]

5. Secondary Outcome: Change in Pain Intensity Score Over 10 Days After Radiotherapy.
Description: Change in pain score over 10 days after radiotherapy, pain score range from 0 (no pain) to 10 (worst pain as can imagine).
Time Frame: Pain intensity score change from baseline of day 0 to day 10 after radiation
Population: Patients with baseline and day 10 pain evaluation.
Measure: Mean (Standard Deviation); unit: units on pain intensity scale
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 130 | 131
units on pain intensity scale | -2.54 (2.88) | -1.99 (2.59)
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Test type: Superiority or Other; p = 0.07, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -0.55, 90% CI 2-sided [-5.06 to 3.97]

ADVERSE EVENTS:
Time Frame: 0 to 6 weeks
Arm/Group | Dexamethasone | Placebo
All-Cause Mortality (participants affected / at risk) | 119/147 | 117/143
Serious Adverse Events (participants affected / at risk) | 0/147 | 0/143
Other Adverse Events (participants affected / at risk) | 119/147 | 117/143
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone (N=147) | Placebo (N=143)
Constipation (Gastrointestinal disorders) | 47 | 37
Diarrhea (Gastrointestinal disorders) | 7 | 10
Dyspepsia (Gastrointestinal disorders) | 12 | 8
Nausea (Gastrointestinal disorders) | 34 | 34
Vomiting (Gastrointestinal disorders) | 9 | 8
Edema limbs (General disorders) | 5 | 8
Fatigue (General disorders) | 58 | 49
Cholesterol high (Investigations) | 8 | 6
Anorexia (Metabolism and nutrition disorders) | 15 | 13
Bone pain (Musculoskeletal and connective tissue disorders) | 61 | 68
Headache (Nervous system disorders) | 9 | 11
Anxiety (Psychiatric disorders) | 11 | 9
Insomnia (Psychiatric disorders) | 26 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 20 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No